CLINICAL TRIAL: NCT02287480
Title: A Phase I/II Dose-finding Randomized, Single-center, Double-blind, Placebo-controlled Safety and Immunogenicity Trial of the Vesicular Stomatitis Virus-vectored Zaire Ebola Candidate Vaccine BPSC1001 (VSVΔG-ZEBOV) in Healthy Adults.
Brief Title: VSV-ZEBOV Geneva Vaccine Trial
Acronym: VSV-ZEBOV
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University Hospital, Geneva (Other)
Collaborators: World Health Organization (Other); Wellcome Trust (Other); Universitätsklinikum Hamburg-Eppendorf (Other); Philipps University Marburg (Other); Albert Schweitzer Hospital (Other); Institute of Tropical Medicine, University of Tuebingen (Other); KEMRI-Wellcome Trust Collaborative Research Program (Other)
Responsible Party: Principal Investigator, Siegrist Claire-Anne, Director of Center for Vaccinology, University Hospital, Geneva
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CCER 14-221
Record Dates: First submitted 2014-11-02; First posted 2014-11-10 (Estimated); Results first posted 2023-05-10 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Ebolavirus Disease
Keywords: Ebolavirus Vaccines

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- VSV-ZEBOV lower dose (Experimental): One intramuscular (deltoid) injection of a lower dose (10^7 plaque-forming units) of VSV-ZEBOV.
  Study amendment (01.2015) : One intramuscular (deltoid) injection of a markedly lower dose (3x 10^5 plaque-forming units) of VSV-ZEBOV
  Interventions: Biological: VSV-ZEBOV
- VSV-ZEBOV higher dose (Experimental): One intramuscular (deltoid) injection of a higher dose (5 x 10^7 pfu) of VSV-ZEBOV.
  Study amendment (01.2015) : interrupted
  Interventions: Biological: VSV-ZEBOV
- Placebo (Placebo Comparator): One intramuscular (deltoid) injection of normal saline (0.5 ml)
  Interventions: Biological: VSV-ZEBOV

INTERVENTIONS:
Biological: VSV-ZEBOV — See arm/group descriptions.
  Other Names: BPSC1001

SUMMARY:
The hemorrhagic fever resulting from Ebola infection is frequently fatal; the current Ebola outbreak, still in its ascendant phase, has a mortality rate over 50%. There is no proven therapy or prevention available at this time.

The vaccine candidate VSV-ZEBOV (BPSC1001) has shown promising safety and efficacy in preventing Ebola Zaire infections in non-human primates (NHP). Before it can be assessed in large Phase IIb/3 trials in affected areas, safety data from phase 1 first-in-human trials are needed. To accelerate this process, the World Health Organization (WHO) has constituted a consortium of Clinical Research Centers in Switzerland, Germany, and Africa that will use similar protocols to collectively include roughly 250 volunteers, the sample size required to identify a 2-fold difference in anti-ZEBOV IgG antibody titers following immunization with 2 different doses of BPSC1001.

The joint primary objectives of this single-center, double-blind, randomized placebo-controlled phase 1 dose-finding study are to assess the safety and tolerability of the VSV-ZEBOV vaccine when administered to healthy volunteers at a lower or higher vaccine dose and to define whether seroresponses differ significantly following immunization with the lower or higher vaccine dose.

DETAILED DESCRIPTION:
This single-center, double-blind, randomized placebo-controlled phase 1 dose-finding study will have two randomization schemes. Volunteers who could later be exposed to Ebolavirus while working in epidemic areas ("deployable subjects") will be randomized to receive one of two vaccine doses. Non-deployable volunteers, with no identified risk of Ebola exposure in the near term, will be allocated to one of three groups and receive the lower or higher vaccine dose, or a placebo. A single immunization will be performed. All subjects will be observed in the clinical trials unit (CTU) for 1.5 hours after vaccine/placebo injection. Subjects will complete post-injection diaries for 7 days after injection, as well as post-injection follow-up visits (see below). On-site visits at the CTU will occur on days -90 to -1, 0, 1, 3, 7, 14, 28, 84, 168. Some subjects with a positive serologic response at 24 weeks may be requested to return for immune durability testing at 12 months.

One or more interim analyses will be undertaken to guide decisions on 1) the potential use of the vaccine in Ph2/3 trials in affected countries and 2) potential modification of the trial(s) through an amendment to evaluate a higher dose, if immunogenicity is poor, or a lower dose if the dosage levels selected are not safe and reasonably well tolerated.

ELIGIBILITY:
Inclusion Criteria:

* Has provided written informed consent before screening
* Adult male or non-pregnant, non-lactating female, ages 18 to 65 (inclusive) at the time of screening
* Free of clinically significant health problems, as determined by pertinent medical history and clinical examination at study screening
* Females of childbearing potential who are willing to use an effective method of contraception, from at least 7 days prior to vaccination through the end of the study period, and a double method from day 0 through day 28
* Males who are willing to use effective contraception from day 0 through day 28:
* Be willing to minimize blood and body fluid exposure of others for 7 days after vaccination
* Use of effective barrier prophylaxis, such as latex condoms, during penetrative sexual intercourse (avoiding the sharing of needles, razors, or toothbrushes, avoiding open-mouth kissing, be willing to refrain from blood donation during the course of the study)

Exclusion Criteria:

* Prior receipt of an Ebolavirus or Marburgvirus vaccine, a VSV-vectored vaccine, or any other investigational vaccine likely to impact on interpretation of the trial data
* Serologic evidence of prior Ebola exposure
* Has a household contact (HHC) who is immunodeficient, HIV-positive, pregnant, has an unstable medical condition in the opinion of the investigator (e.g., New York Heart Association Class ≥ II heart failure, severe debilitating asthma and/or chronic obstructive pulmonary disease)
* Works with livestock
* History of severe local or systemic reactions to any vaccination or a history of severe allergic reactions
* Known allergy to the components of the BPSC1001 vaccine product
* Receipt of investigational product up to 30 days prior to enrollment or ongoing participation in another interventional clinical trial
* Receipt of licensed vaccines within 14 days of planned study immunization (30 days for live vaccines) or ongoing participation in another clinical interventional trial
* Acute or chronic, clinically significant psychiatric, hematologic, pulmonary, cardiovascular, or hepatic or renal functional abnormality as determined by the Investigator based on medical history, physical exam, and/or laboratory screening test
* Any baseline laboratory screening tests which is outside of acceptable range as defined in the protocol: ALT, AST, creatinine, hemoglobin, platelet count, total white blood cell count, urine protein, urine occult blood, urine glucose
* Serologic evidence of hepatitis C infection, evidence of active hepatitis B infection
* Any confirmed or suspected immunosuppressive or immunodeficient condition, including human immunodeficiency virus (HIV) infection, asplenia, cytotoxic therapy in the previous 5 years, and/or diabetes
* Any chronic or active neurologic disorder, including seizures, and epilepsy, excluding febrile seizures as a child
* Has a known history of Guillain-Barré Syndrome
* Has an active malignancy or recent (< 10 years) history of metastatic or hematologic malignancy
* Suspected or known alcohol and/or illicit drug abuse within the past 5 years
* Pregnant or lactating female, or female who intends to become pregnant during the study period
* Administration of immunoglobulins and/or any blood products within the 120 days preceding study entry or planned administration during the study period
* History of blood donation within 30 days of enrollment or plans to donate within the study period
* Administration of chronic (> 14 days) immunosuppressants or other immune-modifying drugs within 6 months of study entry
* Any other significant finding that, in the opinion of the investigator, would increase the risk of the individual's having an adverse outcome by participating in this study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 115 (Actual)
Dates: Start 2014-11; Primary Completion 2015-04 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Claire-Anne Siegrist, MD, Principal Investigator — University Hospita, Geneva
Locations (1):
- University Hospitals of Geneva, Geneva, Switzerland

REFERENCES:
- [Result] Agnandji ST, Huttner A, Zinser ME, Njuguna P, Dahlke C, Fernandes JF, Yerly S, Dayer JA, Kraehling V, Kasonta R, Adegnika AA, Altfeld M, Auderset F, Bache EB, Biedenkopf N, Borregaard S, Brosnahan JS, Burrow R, Combescure C, Desmeules J, Eickmann M, Fehling SK, Finckh A, Goncalves AR, Grobusch MP, Hooper J, Jambrecina A, Kabwende AL, Kaya G, Kimani D, Lell B, Lemaitre B, Lohse AW, Massinga-Loembe M, Matthey A, Mordmuller B, Nolting A, Ogwang C, Ramharter M, Schmidt-Chanasit J, Schmiedel S, Silvera P, Stahl FR, Staines HM, Strecker T, Stubbe HC, Tsofa B, Zaki S, Fast P, Moorthy V, Kaiser L, Krishna S, Becker S, Kieny MP, Bejon P, Kremsner PG, Addo MM, Siegrist CA. Phase 1 Trials of rVSV Ebola Vaccine in Africa and Europe. N Engl J Med. 2016 Apr 28;374(17):1647-60. doi: 10.1056/NEJMoa1502924. Epub 2015 Apr 1. PMID 25830326
- [Result] Huttner A, Dayer JA, Yerly S, Combescure C, Auderset F, Desmeules J, Eickmann M, Finckh A, Goncalves AR, Hooper JW, Kaya G, Krahling V, Kwilas S, Lemaitre B, Matthey A, Silvera P, Becker S, Fast PE, Moorthy V, Kieny MP, Kaiser L, Siegrist CA; VSV-Ebola Consortium. The effect of dose on the safety and immunogenicity of the VSV Ebola candidate vaccine: a randomised double-blind, placebo-controlled phase 1/2 trial. Lancet Infect Dis. 2015 Oct;15(10):1156-1166. doi: 10.1016/S1473-3099(15)00154-1. Epub 2015 Aug 4. PMID 26248510
- [Derived] Huttner A, Agnandji ST, Combescure C, Fernandes JF, Bache EB, Kabwende L, Ndungu FM, Brosnahan J, Monath TP, Lemaitre B, Grillet S, Botto M, Engler O, Portmann J, Siegrist D, Bejon P, Silvera P, Kremsner P, Siegrist CA; VEBCON; VSV-EBOVAC; VSV-EBOPLUS Consortia. Determinants of antibody persistence across doses and continents after single-dose rVSV-ZEBOV vaccination for Ebola virus disease: an observational cohort study. Lancet Infect Dis. 2018 Jul;18(7):738-748. doi: 10.1016/S1473-3099(18)30165-8. Epub 2018 Apr 5. PMID 29627147
- [Derived] Coller BG, Blue J, Das R, Dubey S, Finelli L, Gupta S, Helmond F, Grant-Klein RJ, Liu K, Simon J, Troth S, VanRheenen S, Waterbury J, Wivel A, Wolf J, Heppner DG, Kemp T, Nichols R, Monath TP. Clinical development of a recombinant Ebola vaccine in the midst of an unprecedented epidemic. Vaccine. 2017 Aug 16;35(35 Pt A):4465-4469. doi: 10.1016/j.vaccine.2017.05.097. Epub 2017 Jun 21. PMID 28647166
- [Derived] Medaglini D, Harandi AM, Ottenhoff TH, Siegrist CA; VSV-Ebovac Consortium. Ebola vaccine R&D: Filling the knowledge gaps. Sci Transl Med. 2015 Dec 9;7(317):317ps24. doi: 10.1126/scitranslmed.aad3106. PMID 26659569

RESULTS

PARTICIPANT FLOW:
Groups:
- VSV-ZEBOV High Dose: One intramuscular (deltoid) injection of a "high" dose (10^7 plaque-forming units) of VSV-ZEBOV.
  VSV-ZEBOV: See arm/group descriptions.
- VSV-ZEBOV Highest Dose: One intramuscular (deltoid) injection of a "highest" dose (5 x 10^7 pfu) of VSV-ZEBOV.
  VSV-ZEBOV: See arm/group descriptions.
- VSV-ZEBOV Lowest Dose: Study amendment (01.2015) : One intramuscular (deltoid) injection of a markedly lower dose (3x 10^5 plaque-forming units) of VSV-ZEBOV
Period: Overall Study
Arm/Group | VSV-ZEBOV High Dose | VSV-ZEBOV Highest Dose | Placebo | VSV-ZEBOV Lowest Dose
Started | 35 | 16 | 13 | 51
Completed | 35 | 16 | 13 | 51
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | VSV-ZEBOV High Dose | VSV-ZEBOV Highest Dose | Placebo | VSV-ZEBOV Lowest Dose | Total
Number analyzed (Participants) | 35 | 16 | 13 | 51 | 115
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 44 [34 to 51] | 39 [30 to 54] | 39 [30 to 51] | 40 [29 to 49] | 41 [31 to 51]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 4 | 7 | 27 | 53
  Male | 20 | 12 | 6 | 24 | 62
Region of Enrollment [Number; unit: participants]
  Switzerland | 35 | 16 | 13 | 51 | 115

OUTCOME MEASURES:

1. Primary Outcome: Titers of ZEBOV-specific IgG Antibodies
Description: Primary immunogenicity outcome (required for dose selection)
Time Frame: Day 0 - 28
Population: Note that for many analyses, volunteers vaccinated with either 10^7 or 5x 10^7 pfu were grouped together, as these doses were indistinguishable in immunogenicity and safety profile; see Huttner et al. Lancet Infectious Diseases 2015, Agnandji et al., NEJM 2016.
Measure: Geometric Mean (95% Confidence Interval); unit: ELISA units per ml
Groups:
- VSV-ZEBOV 5x 10^7 OR 10^7 Pfu/ml Dose: Volunteers vaccinated with a single intramuscular (deltoid) injection of either 5x 10^7 plaque-forming units/ml of VSV-ZEBOV or 10^7 pfu/ml of VSV-ZEBOV.
  Note that these two doses proved to be indistinguishable in terms of safety profile and immunogenicity, so the groups were combined for results reporting.
- VSV-ZEBOV 3x 10^5 Pfu/ml Dose: One intramuscular injection (deltoid) of 3x 10^5 pfu/ml of VSV-ZEBOV.
Arm/Group | VSV-ZEBOV 5x 10^7 OR 10^7 Pfu/ml Dose | Placebo | VSV-ZEBOV 3x 10^5 Pfu/ml Dose
Number analyzed (Participants) | 47 | 13 | 51
ELISA units per ml | 1227 [917.3 to 1641.2] | 25 [25.0 to 25.0] | 344.5 [229.7 to 516.4]

2. Secondary Outcome: Number of Participants With Solicited Local and Systemic Reactogenicity Signs and Symptoms
Description: Number of participants with solicited local and systemic reactogenicity signs and symptoms. Day 0 is the day of the study intervention.
Time Frame: Days 0 - 14
Measure: Number; unit: participants
Groups:
- VSV-ZEBOV 5x 10^7 Pfu/ml OR 10^7 Pfu/ml: Volunteers vaccinated with a single intramuscular (deltoid) injection of either 5x 10^7 plaque-forming units/ml of VSV-ZEBOV or 10^7 pfu/ml of VSV-ZEBOV.
  Note that these two doses proved to be indistinguishable in terms of safety profile and immunogenicity, so the groups were combined for results reporting.
- Placebo: volunteers injected with placebo
- Lower Dose (3x10^5 Pfu): Volunteers vaccinated with 3x 10^5 pfu
Arm/Group | VSV-ZEBOV 5x 10^7 Pfu/ml OR 10^7 Pfu/ml | Placebo | Lower Dose (3x10^5 Pfu)
Number analyzed (Participants) | 51 | 13 | 51
participants
  Erythema | 1 | 0 | 0
  Swelling/induration | 2 | 0 | 1
  Pain at injection site | 23 | 3 | 9
  Objective fever | 10 | 0 | 1
  Subjective fever | 20 | 2 | 7
  Chills | 19 | 2 | 14
  Myalgia | 22 | 3 | 14
  Headache | 19 | 4 | 12
  Fatigue | 20 | 4 | 24
  Arthralgia | 6 | 1 | 5

3. Secondary Outcome: Number of Participants With Unsolicited Adverse Events
Description: Number of participants with unsolicited adverse events in the 28 days following injection
Time Frame: Days 0 - 28
Measure: Count of Participants; unit: Participants
Arm/Group | VSV-ZEBOV 5x 10^7 Pfu/ml OR 10^7 Pfu/ml | Placebo | Lower Dose (3x10^5 Pfu)
Number analyzed (Participants) | 51 | 13 | 51
Participants | 11 | 0 | 13

4. Secondary Outcome: Number of Participants With a Serious Adverse Event (SAE)
Description: Number of participants with a serious adverse event (SAE) in the 365 days (1 year) following injection.
Time Frame: Days 0 - 365
Measure: Number; unit: number of participants
Arm/Group | VSV-ZEBOV 5x 10^7 Pfu/ml OR 10^7 Pfu/ml | Placebo | Lower Dose (3x10^5 Pfu)
Number analyzed (Participants) | 51 | 13 | 51
number of participants | 1 | 0 | 1

5. Secondary Outcome: Magnitude (Copies/ml) of VSVΔG-ZEBOV Viremia
Description: Magnitude (copies/ml) of VSVΔG-ZEBOV viremia as expressed by median VSV RNA concentrations after vaccination.
Time Frame: Days 1, 3 and 7
Population: (Note that viremia data for placebo recipients is not reported because these recipients never received vaccine, were never viremic, and thus these data were not collected in these participants.)
Measure: Median (Inter-Quartile Range); unit: VSV RNA copies/ml
Arm/Group | VSV-ZEBOV 5x 10^7 Pfu/ml OR 10^7 Pfu/ml | Lower Dose (3x10^5 Pfu)
Number analyzed (Participants) | 51 | 51
VSV RNA copies/ml
  VSV viremia, day 1 | 323 [65 to 912] | 15 [15 to 15]
  VSV viremia, day 3 (±1) | 178 [65 to 676] | 15 [15 to 15]
  VSV viremia, day 7 (±1) | 15 [15 to 15] | 15 [15 to 15]

6. Secondary Outcome: Persistence of Titers of ZEBOV-specific IgG Antibodies
Description: The percentage of participants maintaining positive ZEBOV-specific IgG antibody titers at 168 days after vaccination.
Time Frame: Day 168
Measure: Count of Participants; unit: Participants
Arm/Group | VSV-ZEBOV 5x 10^7 Pfu/ml OR 10^7 Pfu/ml | Placebo | Lower Dose (3x10^5 Pfu)
Number analyzed (Participants) | 51 | 13 | 51
Participants | 51 | 0 | 49

7. Secondary Outcome: Titers of Neutralizing ZEBOV-specific IgG Antibodies
Description: Geometric mean titers of neutralizing ZEBOV-specific IgG antibodies.
Time Frame: Days 0, 28 and 168
Population: Note that data were ultimately not collected for days 7 and 14.
Measure: Geometric Mean (95% Confidence Interval); unit: Geometric mean titer
Groups:
- VSV-ZEBOV 10^7 Pfu Dose: One intramuscular (deltoid) injection of a lower dose (10^7 plaque-forming units) of VSV-ZEBOV.
  VSV-ZEBOV: See arm/group descriptions.
- VSV-ZEBOV 5x10'^7 Dose: One intramuscular (deltoid) injection of a higher dose (5 x 10^7 pfu) of VSV-ZEBOV.
  Study amendment (01.2015) : interrupted
  VSV-ZEBOV: See arm/group descriptions.
- VSV-ZEBOV 3x10^5 Pfu Dose: Study amendment (01.2015) : One intramuscular (deltoid) injection of a markedly lower dose (3x 10^5 plaque-forming units) of VSV-ZEBOV
Arm/Group | VSV-ZEBOV 10^7 Pfu Dose | VSV-ZEBOV 5x10'^7 Dose | Placebo | VSV-ZEBOV 3x10^5 Pfu Dose
Number analyzed (Participants) | 35 | 15 | 13 | 51
Geometric mean titer
  GMT, day 0 | 4.24 [3.91 to 4.57] | 4.00 [4.00 to 4.00] | 4.00 [4.00 to 4.00] | 4.22 [4.03 to 4.41]
  GMT, day 28 | 13.24 [8.84 to 17.64] | 16.02 [10.23 to 21.81] | 4.11 [3.95 to 4.26] | 14.79 [11.55 to 18.02]
  GMT, day 168 | 7.23 [5.72 to 8.74] | 5.86 [4.49 to 7.23] | 4.54 [4.08 to 4.99] | 6.12 [5.39 to 6.85]

8. Secondary Outcome: Duration of VSVΔG-ZEBOV Viremia
Description: Percentage of participants with any detectable viremia on days 1, 3 and 7
Time Frame: Days 1, 3 and 7
Measure: Count of Participants; unit: Participants
Arm/Group | VSV-ZEBOV 5x 10^7 Pfu/ml OR 10^7 Pfu/ml | Lower Dose (3x10^5 Pfu)
Number analyzed (Participants) | 51 | 51
Participants
  day 1 | 42 | 6
  day 3 | 39 | 8
  day 7 | 1 | 1

9. Secondary Outcome: Number of Participants in Whom Shedding of VSVΔG-ZEBOV Was Detected in Urine and/or Saliva.
Description: This outcome was evaluated in a subset of vaccinees.
Time Frame: Days 1, 3 and 7
Population: Participants in whom shedding of vaccine virus (VSV) was detected in urine or saliva.
Measure: Count of Participants; unit: Participants
Arm/Group | VSV-ZEBOV 5x 10^7 Pfu/ml OR 10^7 Pfu/ml | Placebo | Lower Dose (3x10^5 Pfu)
Number analyzed (Participants) | 30 | 5 | 0
Participants | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Non-serious adverse events were collected in the first 28 days. (Serious adverse events were collected throughout the entire study period, an average of 1 year.)
Arm/Group | VSV-ZEBOV 10^7 Pfu Dose | VSV-ZEBOV 5x10'^7 Dose | Placebo | VSV-ZEBOV 3x10^5 Pfu Dose
Serious Adverse Events (participants affected / at risk) | 1/35 | 0/16 | 0/13 | 1/51
Other Adverse Events (participants affected / at risk) | 8/35 | 3/16 | 0/13 | 13/51
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | VSV-ZEBOV 10^7 Pfu Dose (N=35) | VSV-ZEBOV 5x10'^7 Dose (N=16) | Placebo (N=13) | VSV-ZEBOV 3x10^5 Pfu Dose (N=51)
Hospitalization for left ulnar fracture after a fall (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Left ulnar fracture after a fall, leading to hospitalization for surgical repair. Event considered to have no relationship to the study product.
Hospitalization for rupture of the right quadriceps tendon after a fall (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Volunteer fell while at work. MRI revealed a high-grade rupture of the right quadriceps tendon. Volunteer admitted to the hospital for surgery for debridement and reintegration of the ruptured tendon.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | VSV-ZEBOV 10^7 Pfu Dose (N=35) | VSV-ZEBOV 5x10'^7 Dose (N=16) | Placebo (N=13) | VSV-ZEBOV 3x10^5 Pfu Dose (N=51)
arthritis (Musculoskeletal and connective tissue disorders) | 8 (8) | 3 (3) | 0 (0) | 13 (13) — vaccine-associated arthritis

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes